CLINICAL TRIAL: NCT01956578
Title: REVEAL for Respiration Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REST
Record Dates: First submitted 2013-09-18; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Unexplained Syncope; Suspected Arrhythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breathing Exercise Cohort (Experimental): All patients enrolled will be asked to wear an external respiration band while performing a series of breathing exercises.
  Interventions: Other: Breathing Exercise Cohort

INTERVENTIONS:
Other: Breathing Exercise Cohort — All patients enrolled will be asked to wear a respiration band and perform a series of breathing exercises.

SUMMARY:
This study will evaluate the correlation between the respiratory rate derived from the Reveal Insertable Cardiac Monitor (ICM) electrocardiogram (ECG) with the respiratory rate obtained from an external respiratory band in patients previously implanted with a Reveal for unexplained syncope or suspected arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Subject is implanted with a Reveal ICM or Reveal XT ICM for unexplained syncope or suspected arrhythmia
* Subject (or the legal representative) is willing to sign informed consent form
* Subject is 18 years or older or as specified minimal age per local law/regulation

Exclusion Criteria:

* Significant respiratory diseases such as COPD or pulmonary hypertension.
* Patients with frequent arrhythmias, including PVC's.
* Patients with known heart failure.
* Body conditions that would complicate accurate measurement of respiratory rate with the respiration device.
* Patients which are not able to take the postures as necessary for the study protocol and which cannot walk continuously for a period of 6 minutes.
* Pregnant or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control.
* Subject is enrolled in one or more concurrent studies that would confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Respiration rate derived from the Reveal ICM ECG correlated with the respiration rate from the external respiratory band during a three minute period of normal breathing. | Up to 3 minutes

SECONDARY OUTCOMES:
Respiration rate obtained from the REVEAL ICM ECG with the respiratory rate obtained from external respiratory band during three minute periods of periodic, controlled breathing and elevated heart rate. | Up to 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: J. Bucx, Principal Investigator — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis, Utrecht, Netherlands